CLINICAL TRIAL: NCT02352545
Title: Montelukast for Postinfectious Cough in Adults
Brief Title: Montelukast for Postinfectious Cough
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Liu Min, Beijing Chao Yang Hospital, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Cough
Record Dates: First submitted 2015-01-16; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Cough
MeSH Terms: conditions — Cough | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental: Montelukast (Experimental): Patients in experimental treatment arm were given Montelukast Sodium Tablets (p.o., 10mg, q.d.) .All treatment regimens lasted for 10 days and no other antitussive/decongestant or bronchodilators are given to any patients.
  Interventions: Drug: Montelukast
- Placebo Comparator (Placebo Comparator): Patients in placebo treatment arm were given placebo tablets(main excipient lactose monohydrate,p.o., 10mg, q.d.). All treatment regimens lasted for 10 days and no other antitussive/decongestant or bronchodilators are given to any patients.

INTERVENTIONS:
Drug: Montelukast — Patients in experimental treatment arm were given Montelukast Sodium Tablets (p.o., 10mg, q.d.) .
  Arms: Experimental: Montelukast

SUMMARY:
Cough is a common symptom of respiratory medicine clinic patients, which has complex etiology and wide-ranging. Cough is usually divided into three categories by time: acute cough, subacute cough and chronic cough. Subacute has a 3~8 weeks course of disease. Its main etiology is postinfectious cough, which is mostly secondary to viral infection.Considering its overexpression in postinfectious patient, Cysteinyl leukotriene (CysLTs) plays a role in gathering eosinophils to respiratory. The level of FENO has a significant correlation with inflammatory airway eosinophils. While CysLTs overexpressed in vivo, the level of FENO may increase. Montelukast, as CysLTs-receptor-1 antagonists， plays a role of controlling airway inflammation and decrease airway high activity by suppressing the biological activity of CysLTs. It is effective in theory to therapy sub-acute cough by Montelukast, to short the course and to relieve cough symptoms as soon as possible. The aim is to research whether FENO can be used as a biomarker to optimized treatment regimen of sub-acute cough.

DETAILED DESCRIPTION:
Patients in electrical treatment arm were given Montelukast Sodium Tablets (p.o., 10mg, q.d.) . Patients in placebo treatment arm were given placebo tablets(main excipient lactose monohydrate,p.o., 10mg, q.d.).All treatment regimens lasted for 10 days and no other antitussive/decongestant or bronchodilators are given to any patients.

ELIGIBILITY:
Inclusion Criteria:

* Cough is the main or only clinical symptom and was persistent for 3-8 weeks
* Chest X-ray reveals no noticeable pathological changes

  * 18 year old, regardless of gender and ethical background
* Not taking angiotensin-converting enzyme inhibitor
* Patients must join the programme voluntarily and are able to attend examination and follow-up sessions

Exclusion Criteria:

* Patients diagnosed with allergic rhinitis, chronic nasosinusitis or bacterial respiratory tract infections
* Patients diagnosed with severe reportorial disease of other severe systemic disease
* Patients who are allergic to any drugs to be tested
* Patients who are non-cooperative during examination sessions or other steps of the trial
* Patients who are not able to or refuse to sign consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Change in Leicester Cough Questionnaire(LCQ) total and domain scores at 10 days post randomisation | 10 days

SECONDARY OUTCOMES:
cough visual analogue scale scores post randomisation(area under the curve) | 10 days
Change in Leicester Cough Questionnaire(LCQ) physical,psychological and social domain scores at 10 days post randomisation | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Kewu Huang, M.D., Study Director — Beijing Chao Yang Hospital
Locations (1):
- Kewu Huang, China, Beijing Municipality, China

REFERENCES:
- [Background] Morice AH, Fontana GA, Sovijarvi AR, Pistolesi M, Chung KF, Widdicombe J, O'Connell F, Geppetti P, Gronke L, De Jongste J, Belvisi M, Dicpinigaitis P, Fischer A, McGarvey L, Fokkens WJ, Kastelik J; ERS Task Force. The diagnosis and management of chronic cough. Eur Respir J. 2004 Sep;24(3):481-92. doi: 10.1183/09031936.04.00027804. No abstract available. PMID 15358710
- [Background] Kwon NH, Oh MJ, Min TH, Lee BJ, Choi DC. Causes and clinical features of subacute cough. Chest. 2006 May;129(5):1142-7. doi: 10.1378/chest.129.5.1142. PMID 16685003
- [Background] McCool FD. Global physiology and pathophysiology of cough: ACCP evidence-based clinical practice guidelines. Chest. 2006 Jan;129(1 Suppl):48S-53S. doi: 10.1378/chest.129.1_suppl.48S. PMID 16428691
- [Background] Mita H, Turikisawa N, Yamada T, Taniguchi M. Quantification of leukotriene B4 glucuronide in human urine. Prostaglandins Other Lipid Mediat. 2007 Feb;83(1-2):42-9. doi: 10.1016/j.prostaglandins.2006.09.010. Epub 2006 Dec 5. PMID 17259071
- [Background] Ryan NM, Gibson PG. Extrathoracic airway hyperresponsiveness as a mechanism of post infectious cough: case report. Cough. 2008 Aug 4;4:7. doi: 10.1186/1745-9974-4-7. PMID 18673583
- [Background] Cho YS, Park SY, Lee CK, Lee EY, Shin JH, Yoo B, Moon HB. Enhanced cough response to hyperpnea with cold air challenge in chronic cough patients showing increased cough sensitivity to inhaled capsaicin. Allergy. 2003 Jun;58(6):486-91. doi: 10.1034/j.1398-9995.2003.00183.x. PMID 12757448
- [Background] Montuschi P, Mondino C, Koch P, Barnes PJ, Ciabattoni G. Effects of a leukotriene receptor antagonist on exhaled leukotriene E4 and prostanoids in children with asthma. J Allergy Clin Immunol. 2006 Aug;118(2):347-53. doi: 10.1016/j.jaci.2006.04.010. Epub 2006 Jul 3. PMID 16890757
- [Background] Kato A, Schleimer RP. Beyond inflammation: airway epithelial cells are at the interface of innate and adaptive immunity. Curr Opin Immunol. 2007 Dec;19(6):711-20. doi: 10.1016/j.coi.2007.08.004. Epub 2007 Oct 24. PMID 17928212
- [Background] Sato S, Saito J, Sato Y, Ishii T, Xintao W, Tanino Y, Ishida T, Munakata M. Clinical usefulness of fractional exhaled nitric oxide for diagnosing prolonged cough. Respir Med. 2008 Oct;102(10):1452-9. doi: 10.1016/j.rmed.2008.04.018. Epub 2008 Jul 9. PMID 18614345
- [Background] Kerr JB. Functional cytology of the human testis. Baillieres Clin Endocrinol Metab. 1992 Apr;6(2):235-50. doi: 10.1016/s0950-351x(05)80149-1. PMID 1616444
- [Background] Seymour ML, Gilby N, Bardin PG, Fraenkel DJ, Sanderson G, Penrose JF, Holgate ST, Johnston SL, Sampson AP. Rhinovirus infection increases 5-lipoxygenase and cyclooxygenase-2 in bronchial biopsy specimens from nonatopic subjects. J Infect Dis. 2002 Feb 15;185(4):540-4. doi: 10.1086/338570. Epub 2002 Jan 31. PMID 11865407
- [Background] Gentile DA, Fireman P, Skoner DP. Elevations of local leukotriene C4 levels during viral upper respiratory tract infections. Ann Allergy Asthma Immunol. 2003 Sep;91(3):270-4. doi: 10.1016/S1081-1206(10)63529-6. PMID 14533659